CLINICAL TRIAL: NCT07292792
Title: Integration of Peer Health Navigation Into Comprehensive Re-entry Services: Improving PrEP Implementation for Justice-involved Individuals
Brief Title: The Unlocking PrEP Study: Integration of Peer Health Navigation Into Comprehensive Re-entry Services
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Unlocking Doors (Unknown)
Responsible Party: Principal Investigator, Ank Nijhawan, Professor- Internal Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0736
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: HIV Disease; HIV Prevention
Keywords: PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Coach Intervention Group: Participants in this group are clients of Unlocking Doors who meet eligibility criteria and choose to enroll in the study. They receive the health coach intervention, which includes general health and sexual health discussions, HIV and syphilis testing, PrEP education, PrEP eligibility screening, linkage to PrEP care, and referrals to other health or re-entry services. Their PrEP knowledge, interest, and engagement, as well as feasibility and acceptability of the model, are assessed throughout the study.
  Interventions: Behavioral: Health Coach Intervention

INTERVENTIONS:
Behavioral: Health Coach Intervention — The intervention integrates a PrEP-focused health coach into Unlocking Doors' re-entry services. The health coach provides clients with general health guidance, sexual health education, HIV and syphilis testing, PrEP education, PrEP eligibility screening, and linkage to PrEP care. The coach also offers ongoing navigation and referrals to medical, behavioral health, and re-entry services as needed. The aim of the intervention is to increase PrEP awareness, interest, and uptake among justice-involved individuals while assessing feasibility, acceptability, and appropriateness of embedding a health coach within legal re-entry services.

SUMMARY:
This 18-month study, "Integration of peer health navigation into comprehensive re-entry services: improving PrEP implementation for justice-involved individuals," aims to increase PrEP awareness and uptake among people with a history of justice involvement in Dallas, primarily clients of Unlocking Doors.

DETAILED DESCRIPTION:
This 18-month study, "Integration of peer health navigation into comprehensive re-entry services: improving PrEP implementation for justice-involved individuals," aims to increase PrEP awareness and uptake among people with a history of justice involvement in Dallas, primarily clients of Unlocking Doors. Guided by the EPIS (Exploration, Preparation, Implementation, Sustainment) framework, the study will:

Conduct qualitative interviews with Unlocking Doors staff, clients, health coaches, and PrEP providers to identify barriers and facilitators to integrating a health coach focused on sexual health, HIV testing, and PrEP.

Use rapid qualitative analysis to adapt the health coach intervention and workflows.

Implement a health coach model embedded in Unlocking Doors to offer general and sexual health discussions, PrEP education, HIV/syphilis testing, and linkage to PrEP care and other services.

Enroll up to 600 consented/screened individuals to achieve a target of 100 participants in the intervention.

Assess feasibility, acceptability, and appropriateness of the model, as well as changes in PrEP knowledge, interest, referrals, and uptake over time.

The study is led by PI: Ank Nijhawan in UTSW Infectious Diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Client of Unlocking Doors
3. Able to provide informed consent
4. Willing to participate in discussions about general health, sexual health, HIV prevention, and PrEP
5. Willing to complete health screening and eligibility assessment
6. For qualitative interview participants:

   * Unlocking Doors staff, clients, or PrEP providers who agree to participate in a one-time interview.

Exclusion Criteria:

1. Under 18 years of age
2. Unable to provide informed consent
3. Not receiving services at Unlocking Doors
4. Non-English speakers
5. Diagnosed with HIV
6. Incarcerated individuals at the time of recruitment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18+) receiving re-entry services at Unlocking Doors, including justice-involved individuals and staff participating in qualitative interviews. Participants are engaged in general health, sexual health, and PrEP-related discussions with a health coach as part of the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Integrating a PrEP-Focused Health Coach | 18 Months
  Feasibility will be assessed by the proportion of Unlocking Doors clients who engage with the health coach. This indicator reflects whether the health coach can be effectively integrated into existing re-entry workflows.
Acceptability of the Health Coach Model | 18 Months
  Acceptability will be assessed using custom questions developed by our team and modified question items from the Scales for Participant Alliance with Recovery Coach (SPARC) scale, and which will be asked of clients and staff. These questions will assess satisfaction, comfort, and perceived usefulness of health coach interactions. Response options will be rated on a Likert scale ranging from 1 - 5, with higher scores indicating better perceptions of acceptability. Qualitative feedback will supplement these ratings to capture overall acceptability.
Appropriateness of the Health Coach Model | 18 Months
  Appropriateness will be assessed using custom questions developed by our team and modified question items from the Scales for Participant Alliance with Recovery Coach (SPARC) scale. These questions assess perceived relevance, fit, and value of integrating a health coach into Unlocking Doors' services, as well as how well the model aligns with client needs. Response options will be rated on a Likert scale ranging from 1 - 5, with higher scores indicating better perceptions of appropriateness. Qualitative feedback will supplement these ratings to capture overall appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Ank E Nijhawan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States